CLINICAL TRIAL: NCT01567371
Title: Use of the LiDCORapid Monitor in Patients During Graded Phlebotomy and the Removal of Autologous Blood
Brief Title: LiDCO Monitor Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Joseph D. Tobias, Chairman, Dept. of Anesthesiology & Pain Medicine, Nationwide Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB12-00096
Record Dates: First submitted 2012-03-26; First posted 2012-03-30 (Estimated); Results first posted 2016-04-15 (Estimated); Last update posted 2016-04-15 (Estimated); Status verified 2016-03

CONDITIONS: Cardiac Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LiDCO rapid monitor (Experimental)
  Interventions: Device: LiDCO rapid monitor

INTERVENTIONS:
Device: LiDCO rapid monitor — Technology which provides a continuous means of monitoring various hemodynamic parameters including cardiac output and pulse pressure variability.

SUMMARY:
This is a study to validate the utility and accuracy of the non-invasive device (LiDCOrapid monitor) during a period of phlebotomy and graded blood loss in patients who are having cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for intraoperative phlebotomy following anesthetic induction to obtain autologous blood for use following cardiopulmonary bypass and cardiac surgery.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-03; Primary Completion 2014-12 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | LiDCO Rapid Monitor
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | LiDCO Rapid Monitor
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 16
  Between 18 and 65 years | 14
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.5 (11.018)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 15
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Difference in Pulse Pressure Variability From Baseline to Post-ANH
Description: The difference in pulse pressure variability during a period of phlebotomy and graded blood loss, measured before phlebotomy or acute normovolemic hemodilution (ANH) and immediately after.
Time Frame: 1 Day
Measure: Mean (Standard Deviation); unit: % variability
Arm/Group | LiDCO Rapid Monitor
Number analyzed (Participants) | 30
% variability | 7.46 (9.149)

2. Secondary Outcome: Difference in Stroke Volume Variability From Baseline to Post ANH.
Description: The difference in stroke volume variability during a period of phlebotomy and graded blood loss, measured before phlebotomy or acute normovolemic hemodilution (ANH) and immediately after.
Time Frame: 1 Day
Measure: Mean (Standard Deviation); unit: % variability
Arm/Group | LiDCO Rapid Monitor
Number analyzed (Participants) | 30
% variability | 4.46 (5.368)

ADVERSE EVENTS:
Arm/Group | LiDCO Rapid Monitor
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes